CLINICAL TRIAL: NCT06602635
Title: A Hybrid Score to Predict the Origin of Outflow Tract Ventricular Arrhythmias in Patients with Intraventricular Conduction Disorders or Paced Rhythm
Brief Title: Hybrid Score to Predict OTVA-SOO in Patients with Wide Basal QRS
Status: Recruiting | Type: Observational
Sponsor: Centro Medico Teknon (Other)
Collaborators: Hospital Universitario Puerta del Mar (Other); Vrije Universiteit Brussel (Other); Cisanello University Hospital (Pisa, Italy) (Unknown); Maria Cecilia Hospital (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, MD, PhD, Centro Medico Teknon
Other Study IDs: Hybrid-score OTVA
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: ECG; Ventricular Arrhythmias; Catheter Ablation
Keywords: Ventricular extrasystole; Premature ventricular complex; ecg; outflow tract ventricular arrhythmias
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RVOT origin: Patients with right ventricular outflow tract (RVOT) arrhythmias origin
  Interventions: Diagnostic Test: ECG and clinical score
- LVOT origin: Patients with left ventricular outflow tract (LVOT) arrhythmias origin
  Interventions: Diagnostic Test: ECG and clinical score

INTERVENTIONS:
Diagnostic Test: ECG and clinical score — The Hybrid Score (HS), detailed in previous literature involves a sum of points based on clinical and ECG characteristics. Points are assigned as follows: one point each for being over 50 years old, male, and having arterial hypertension. ECG-based points are allocated according to QRS transition: 3 points for a transition in V1, 2 points for V2, 1 point for V3 if the R-wave in V3 is greater than 1 mV; 1 point is subtracted if V3 has an R-wave less than 1 mV, and further deductions or additions apply for transitions up to V6. A score ≤ 1 suggests an RVOT origin, whereas ≥ 2 suggests an LVOT origin.

SUMMARY:
Outflow tract ventricular arrhythmia (OTVA) is the most common type of ventricular arrhythmia, and catheter ablation (CA) is the primary treatment option for patients experiencing symptoms. Accurately identifying the origin site of OTVA is essential for effective catheter ablation, minimizing procedural risks, and enhancing treatment success. However, most studies that developed algorithms or scoring systems for distinguishing OTVA origins excluded participants with structural heart disease and those with paced rhythms from their study groups. A recent prospective evaluation of a hybrid score (HS) that integrates both clinical and ECG data to predict OTVA-SOO, including patients with cardiac implantable electronic devices and those with structural heart disease in our study.

The presented study aimed to assess the effectiveness of the previously described hybrid algorithm in predicting OTVA-SOO in a patient population characterized by a wide basal QRS due to intraventricular conduction defects or paced rhythms.

The Hybrid Score The Hybrid Score (HS), involves a sum of points based on clinical and ECG characteristics. Points are assigned as follows: one point each for being over 50 years old, male, and having arterial hypertension. ECG-based points are allocated according to QRS transition: 3 points for a transition in V1, 2 points for V2, 1 point for V3 if the R-wave in V3 is greater than 1 mV; 1 point is subtracted if V3 has an R-wave less than 1 mV, and further deductions or additions apply for transitions up to V6. A score ≤ 1 suggests an RVOT origin, whereas ≥ 2 suggests an LVOT origin.

ECGs were recorded with a standard configuration at a 25 mm/s sweep speed.

Premature Ventricular Contraction (PVC) Ablation Activation mapping of spontaneous OTVAs was conducted. The procedure aimed to abolish spontaneous OTVAs, with the site of ablation marking the site of origin (SOO).

Collected data

* Patient Information and Consent (procedure must be done within 60 days of consent)
* Demographics (age, gender, etc.)
* Vital signs (length, weight, etc.)
* Medical history, including cardiovascular risk factors, cardiomyopathy and drugs
* ECG data
* Echocardiographic data (left ventricular ejection fraction and left ventricular end-diastolic diameter)
* Procedure data (number of radiofrequency applications, site of effective ablation, total radiofrequency time, total fluoro time, points mapping, procedure time)
* Adverse Events

ELIGIBILITY:
Inclusion Criteria:

* ventricular arrhythmia with a morphology indicating an outflow tract origin and a wide basal QRS complex
* a QRS width greater than 110 ms was considered wide
* willing and capable of providing written informed consent to the study

Exclusion Criteria:

* catether ablation procedure was unsuccessful
* infrequent arrhythmia requiring ablation guided by pacemapping.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population undergoing catheter ablation for outflow tract ventricular arrhythmias
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-23 (Estimated)

PRIMARY OUTCOMES:
Hybrid score performance | At the moment of interventional procedure
  The primary endpoint of the study is to establish the sensibility and specificity of an already validated clinical and electrocardiographic score for the prediction of left or right outflow tract ventricular arrhythmias in a selected population with large QRS because of intraventricular conduction disorders or paced rhythm who underwent catheter ablation of the arrhythmia.

SECONDARY OUTCOMES:
Safety | 1 month after the procedure date
  The safety outcome is the incidence of post-procedural major adverse events

CONTACTS AND LOCATIONS:
Locations (6):
- Vrije Universiteit Brussel, Brussels, Belgium, Belgium
- Italy (3):
  - Maria Cecilia Hospital, Cotignola, Italy
  - Niguarda Ca Granda Hospital, Milan, Italy
  - Cisanello University Hospital (Pisa, Italy), Pisa, Italy
- Spain (2):
  - Teknon Medical Center, Barcelona, Spain
  - Hospital Universitario Puerta del Mar, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeppenfeld K, Tfelt-Hansen J, de Riva M, Winkel BG, Behr ER, Blom NA, Charron P, Corrado D, Dagres N, de Chillou C, Eckardt L, Friede T, Haugaa KH, Hocini M, Lambiase PD, Marijon E, Merino JL, Peichl P, Priori SG, Reichlin T, Schulz-Menger J, Sticherling C, Tzeis S, Verstrael A, Volterrani M; ESC Scientific Document Group. 2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. Eur Heart J. 2022 Oct 21;43(40):3997-4126. doi: 10.1093/eurheartj/ehac262. No abstract available. PMID 36017572
- [Background] Anderson RD, Kumar S, Parameswaran R, Wong G, Voskoboinik A, Sugumar H, Watts T, Sparks PB, Morton JB, McLellan A, Kistler PM, Kalman J, Lee G. Differentiating Right- and Left-Sided Outflow Tract Ventricular Arrhythmias: Classical ECG Signatures and Prediction Algorithms. Circ Arrhythm Electrophysiol. 2019 Jun;12(6):e007392. doi: 10.1161/CIRCEP.119.007392. Epub 2019 Jun 4. PMID 31159581